CLINICAL TRIAL: NCT02650609
Title: Treatment of Chronic Subdural Hematoma by Corticosteroids
Acronym: SUCRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-000927-96
Record Dates: First submitted 2016-01-04; First posted 2016-01-08 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Chronic Subdural Hematomas
Keywords: chronic subdural hematomas; surgical treatment; corticosteroids
MeSH Terms: conditions — Hematoma, Subdural, Chronic | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methylprednisolone (Experimental): Methylprednisolone will be supplied as powder and stored in capsules containing 16 mg with lactose as excipient.
  Capsules will be administered orally in the morning, during breakfast with a glass of water.
  Dose is adapted according to the weight of the patient (1mg/kg):
  * <60 kg: 3 pills of 16 mg/day
  * 60-80kg: 4 pills of 16 mg/day
  * >80kg: 5 pills of 16 mg/day The duration of the treatment is 21 days.
  Interventions: Drug: Methylprednisolone
- Placebo (Placebo Comparator): Placebo capsules will only contain lactose. Capsules will be administered orally in the morning, during breakfast with a glass of water.
  Dose is adapted according to the weight of the patient (1mg/kg):
  * <60 kg: 3 pills of 16 mg/day
  * 60-80kg: 4 pills of 16 mg/day
  * >80kg: 5 pills of 16 mg/day The duration of the treatment is 21 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylprednisolone
  Arms: Methylprednisolone
Drug: Placebo
  Arms: Placebo

SUMMARY:
Chronic subdural hematomas are a frequent neurosurgical pathology in the elderly. Gold standard is surgical evacuation of these hematomas. Physiopathology of chronic subdural hematoma involves numerous inflammatory processes which could be inhibited by steroids.

DETAILED DESCRIPTION:
The primary objective is to evaluate the efficacy of corticosteroids treatment in patients with Chronic subdural hematomas without clinical or radiological signs of severity.

Secondary objectives are to assess the effect of methylprednisolone on:

* quality of life evolution,
* morbidity and mortality,
* radiological evolution of the lesions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old,
* With chronic or subacute, uni or bilateral subdural hematoma,
* Confirmed by cerebral scan without contrast enhancement,
* Without clinical and radiological signs of severity,
* Written informed consent from patients or their next of kin according to the patients cognitive status.

Exclusion Criteria:

* Diabetics patients,
* Contraindication for methylprednisolone,
* Previous surgery for chronic subdural hematoma during the past 6 months,
* Pre-existing severe dementia related to other etiology than the Chronic subdural hematomas,
* Existing neurological pathology that can be associated with dementia,
* Patients treated with corticosteroids,
* Protected person (adults legally protected (under judicial protection, guardianship or supervision), person deprived of their liberty, pregnant woman, lactating woman and minor),
* Participating in other concomitant research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2016-06-24 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Delay of occurrence of surgical treatment of the Chronic subdural hematomas | 1 month

SECONDARY OUTCOMES:
Quality of life score | 1, 3 and 6 months
  Short Form Health Survey 12 scale
Time to surgical treatment | during the first 6 months
Rate of surgical treatment of the Chronic subdural hematomas | 1, 3 and 6 months
Functional scales : daily living | 1, 3 and 6 months
  Instrumental Activities of Daily Living scale
Functional scales : cognitive | 1, 3 and 6 months
  Mini-Mental State Examination scale
Functional scales : modified Rankin Scale | 1, 3 and 6 months
  modified Rankin Scale
Plasma sodium | day 0, 7, 14, and 21 and 1 month
Potassium | day 0, 7, 14, and 21 and 1 month
Fasting glucose | day 0, 7, 14, and 21 and 1 month
Occurrence of adverse events potentially related to methylprednisolone | during the first 6 months
Survival | 6 months
Radiological improvement | 1, 3 and 6 months
  Radiological improvement defined by reduction of maximal thickness of hematoma and reduction of midline shift evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Xavier XM MORANDI, MD, PhD, Principal Investigator — CHU Rennes; Pierre-Louis PH HENAUX, MD, Principal Investigator — CHU Rennes; Pierre-Jean PL LE RESTE, MD, Principal Investigator — CHU Rennes
Locations (17):
- France (17):
  - CHU Amiens, Amiens
  - CHU Angers, Angers
  - CHU Besançon, Besançon
  - CHU Bordeaux Neurochirurgie A, Bordeaux
  - CHU Bordeaux Neurochirurgie B, Bordeaux
  - CHU Brest, Brest
  - CHU Caen, Caen
  - CHU Lille, Lille
  - HC Lyon, Lyon
  - AP-HM - Hôpital La Timone, Marseille
  - CHU Nancy, Nancy
  - CHU Nantes, Nantes
  - CHU Poitiers, Poitiers
  - CHU Rouen, Rouen
  - CHU Saint Etienne, Saint-Etienne
  - CHU Strasbourg, Strasbourg
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Henaux PL, Le Reste PJ, Laviolle B, Morandi X. Steroids in chronic subdural hematomas (SUCRE trial): study protocol for a randomized controlled trial. Trials. 2017 Jun 5;18(1):252. doi: 10.1186/s13063-017-1990-8. PMID 28583162